CLINICAL TRIAL: NCT02660151
Title: Prospective, Randomized Crossover Study of Using the Hyper-CL™ Lens (Hyper Osmotic Contact Lens) in Subjects Suffering From Corneal Edema
Brief Title: Study of Using the Hyper-CL™ Lens (Hyper Osmotic Contact Lens) in Subjects Suffering From Corneal Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye-yon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ECL00030
Record Dates: First submitted 2016-01-11; First posted 2016-01-21 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: CORNEAL EDEMA
MeSH Terms: conditions — Corneal Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A-B (Experimental): Treatment A: Hyper-CL™ lens + salt solution + antibiotics drops (7 days) Treatment B: Regular soft contact lens +salt solution+ antibiotics drops (7 days) One week (7 days) of washout without any treatment will be between treatments.
  Interventions: Device: Hyper-CL™ lens; Device: Regular soft contact lens; Drug: Salt solution
- Treatment B-A (Experimental): Treatment A: Hyper-CL™ lens + salt solution + antibiotics drops (7 days) Treatment B: Regular soft contact lens +salt solution+ antibiotics drops (7 days) One week (7 days) of washout without any treatment will be between treatments.
  Interventions: Device: Hyper-CL™ lens; Device: Regular soft contact lens; Drug: Salt solution

INTERVENTIONS:
Device: Hyper-CL™ lens
Device: Regular soft contact lens
Drug: Salt solution

SUMMARY:
The Hyper-CL™ lenses are indicated for therapeutic use as a bandage to protect the corneal surface and to relieve corneal pain in the treatment of acute or chronic ocular pathologies, such as bullous keratopathy, corneal erosions, entropion, corneal edema, and corneal dystrophies as well as post-surgical conditions resulting from cataract extraction and corneal surgery. The lenses may be prescribed for daily wear with removal for cleaning and disinfection (chemical, not heat) prior to reinsertion, as recommended by the eye care professional.

In addition Hyper-CL™ contact lenses can also provide optical correction during healing if required.

DETAILED DESCRIPTION:
This study is a prospective, randomized crossover study. The primary aim of this study is to assess the safety and effectiveness of using the Hyper-CL™ lens +salt solution (5% NaCl) as compared with using regular contact lens + salt solution (5% NaCl) in subjects suffering from corneal edema. Safety will be assessed by evaluating the rate of adverse events and adverse device effects occurred throughout the study period. Effectiveness will be assessed by measuring changes in corneal thickness and visual acuity.

Subjects with corneal edema will be the study population. Only subjects who have signed the informed consent form and meet all the eligibility criteria listed below will be qualified for enrollment. The study will encompass a total of up to 80 subjects who will complete the Protocol follow-up schedule.

Each subject will be treated with:

Treatment A: Hyper-CL™ lens + salt solution + antibiotics drops (7 days) Treatment B: Regular soft contact lens +salt solution+ antibiotics drops (7 days) One week (7 days) of washout without any treatment will be between treatments. Subject will be equally allocated to one of the following 2 crossover regimen based on a randomization scheme with blocks stratified by center: A-B; B-A

ELIGIBILITY:
Inclusion Criteria:

1. Subject is over 18 years old
2. Subject with corneal edema in the visual access
3. Subject with visual acuity of 6/20 or worse (equivalent ETDRS) clinically explained by corneal edema
4. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed.

Exclusion Criteria:

1. Subject with active Herpes keratitis
2. Subject with scarred cornea
3. Subject who is suffering from erosions and/or infections of the cornea (red eye)
4. Subject with glaucoma shunts (e.g. Ahmed valve) and or bleb
5. Subject who require chronic administration of any topical ophthalmic beside lubrication eye drops and steroids or anti glaucoma drags
6. Subject who is currently participating or have participated in an investigational study, other than this study, within the past 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-02; Primary Completion 2018-10 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
frequency and severity of all treatment-related adverse events | Up to 28 days (or 21 days if wash out is not needed).
Percent of subjects with corneal thickness decrease of at least 8% and or visual acuity improvement of at least 1 line following treatment with the Hyper-CL™ lens + salt solution | Up to 28 days (or 21 days if wash out is not needed).
  assess by physiological parameter

SECONDARY OUTCOMES:
Percent of subjects with corneal thickness decrease of at least 8%. | Up to 28 days (or 21 days if wash out is not needed).
  assess by physiological parameter
Percent of subjects with visual acuity improvement of at least 1 line | Up to 28 days (or 21 days if wash out is not needed).
  assess by physiological parameter
Corneal thickness decrease | Up to 28 days (or 21 days if wash out is not needed).
  assess by physiological parameter
change in Measurement Best Corrected Distance Visual Acuity (BCDVA) | Up to 28 days (or 21 days if wash out is not needed).
change in Subject comfort questionnaire | Up to 28 days (or 21 days if wash out is not needed).

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (2):
  - Soroka MC, Beersheba
  - Sheba MC, Ramat Gan
- Poland (2):
  - Katowice MC, Katowice
  - Lublin MC, Lublin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Daphna O, Mimouni M, Keshet Y, Ben Ishai M, Barequet IS, Knyazer B, Mrukwa-Kominek E, Zarnowski T, Chen-Zion M, Marcovich A. Therapeutic HL-Contact Lens versus Standard Bandage Contact Lens for Corneal Edema: A Prospective, Multicenter, Randomized, Crossover Study. J Ophthalmol. 2020 Sep 21;2020:8410920. doi: 10.1155/2020/8410920. eCollection 2020. PMID 33014443